CLINICAL TRIAL: NCT04348344
Title: Study on the Prevention and Control System of Chronic Airway Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hongtao Niu, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-161-K110
Record Dates: First submitted 2020-04-07; First posted 2020-04-16 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; asthma; pulmonary rehabilitation; air pollutans
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): health education of pulmonary rehabilitation pulmonary rehabilitation including aerobic exercise，strength training and breath training.
  Patients in stable stages using the "home-based rehabilitation" exercise prescription, taking home exercise, using the sports bracelet and special respiratory rehabilitation app software, the home management system integrating home rehabilitation training, detection and feedback is mainly adopted, which is a combination of aerobic endurance training, intermittent strength training and inspiratory muscle training.
  Interventions: Behavioral: pulmonary rehabilitation
- control group (No Intervention): health education of pulmonary rehabilitation

INTERVENTIONS:
Behavioral: pulmonary rehabilitation — Patients receive health education of pulmonary rehabilitation, using the "home-based rehabilitation" exercise prescription, taking home exercise as the main form, using the sports bracelet and special respiratory rehabilitation app software, the home management system integrating home rehabilitation training, detection and feedback is mainly adopted, which is a combination of aerobic endurance training: walking, intermittent strength training: elastic band and inspiratory muscle training:apparatus, abdominal breathing training.
  Arms: intervention group

SUMMARY:
In this study, patients with Chronic Obstructive Pulmonary Diseases (COPD) in stable and acute exacerbation stage were selected as the research objects, and the open, parallel and randomized controlled clinical trial design was adopted. Participants were randomly divided into trial group and control group. The control group was only given routine education, and the experimental group, on the basis of routine education, developed a respiratory rehabilitation training program lasting for 12 weeks according to the individual situation of patients. All participants were interviewed for 6 times (baseline and 4,8,12 weeks, 6 months and 12 months after admission) for a period of 1 year. Acute exacerbation, activity tolerance (6-minute walking test), living environment, clinical symptoms, lung function, airway inflammation water level index and biological samples were collected at each visit. At the same time, according to the diary filled in by the patients, the investigators can obtain the daily stay time indoors and outdoors and the longitude and latitude information of the regular stay fixed place, and geographic information system (GIS) is used to match the nearest environmental monitoring station, obtain the data of air pollutants and meteorological indicators (SO2, NO2, Co, O3, PM10, temperature and humidity, etc.), and estimate the individual exposure level of air pollutants.

DETAILED DESCRIPTION:
First of all, the investigators need to obtain detailed history records, including cardio pulmonary vascular history, related complications, treatment history and other high-risk factors. After careful review, the investigators need to determine whether the patient is suitable to participate in the pulmonary rehabilitation plan. The investigators need to pay special attention to diseases that may affect the patient's performance, including special cardiovascular diseases, skeletal muscle and nervous system.

Functional evaluation: pulmonary function test, exercise cardiopulmonary function evaluation (6-minute walking test), grip strength test, psychological state evaluation ( Generalized Anxiety Disorder 7-item (GAD-7), Patient Health Questionnaire 9-item (phq-9)), nutrition screening and evaluation and others (general examination such as height, weight, BMI, waist and hip circumference, WHR, blood pressure, heart rate and blood biochemical examination; quality of life evaluation; other related individual evaluation Estimation includes smoking and sleep).

1. Acute exacerbation:

   The exercise prescription of "hospitalization + home rehabilitation" was adopted, which mainly combined aerobic endurance training, intermittent strength training and inspiratory muscle training, as follows:

   Aerobic exercise: 4 times / week, 30min / time, fast walking or power cycling Strength training: unarmed or instrument, 4 times / week, 3 groups / time, 10-12 times / group Breath training: ① breath Trainer: once a day, 20-30min a time

   ② Abdominal breathing training: 1-2 times / day, 10min / time
2. Stable patients:

Using the "home-based rehabilitation" exercise prescription, taking home exercise as the main form, using the sports bracelet and special respiratory rehabilitation app software, the home management system integrating home rehabilitation training, detection and feedback is mainly adopted, which is a combination of aerobic endurance training, intermittent strength training and inspiratory muscle training, as follows:

Aerobic exercise: 2-3 times / week, 30min / time, walk quickly Strength training: elastic band, 2-3 times / week, 3 groups / time, 10-12 times / group Breathing training: ① breathing exercise apparatus, 1-2 times / day, 10min / time

② Abdominal breathing training, 1-2 times / day, 10min / time

ELIGIBILITY:
Inclusion Criteria:

* It meets the diagnostic criteria of global initiative for chronic obstructive pulmonary disease (gold 2017 Edition), is in a stable period of disease or meets the diagnostic criteria of guidelines for the prevention and treatment of bronchial asthma (GINA 2016 Edition)
* Have lived in the local area for more than 2 consecutive years, and there is no plan to go out for more than half a year in succession during the survey period
* No smoking history or no smoking for half a year or more
* 40-75 years old

Exclusion Criteria:

* Patients with history of chronic diseases, such as serious cardiovascular and cerebrovascular diseases, liver and kidney dysfunction, epilepsy and other nervous system diseases, mental diseases, psychiatric diseases, active pulmonary tuberculosis, tumor, anti tuberculosis treatment or combined influence information collection
* Patients who have undergone thoracic, abdominal and ophthalmic operations in the past 3 months
* Pregnant and lactating women
* Did not sign informed consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline 6-minute Walking Distance at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  walking distance in 6-minute walking test
Times of acute exacerbation | through study completion, an average of 1 year
  times of acute exacerbation in the period of one year

SECONDARY OUTCOMES:
Time from the beginning of follow-up to the first acute exacerbation and the duration of the first acute exacerbation | 9 months
  Time from the beginning of follow-up to the first acute exacerbation and the duration of the first acute exacerbation
Change from Baseline Fractional exhaled Nitric Oxide (FeNO) at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  changes of Fractional exhaled Nitric Oxide (FeNO)
Change from Baseline Eosinophil Count in Sputum at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  Eosinophil Count
Change from Baseline Inflammatory Factors in sputum at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  inflammatory factors in sputum
Change from Baseline modified Medical Research Council dyspnea (mMRC) at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  the minimum values is 0 and maximum values is 4, the higher scores mean a worse outcome.
Change from Baseline COPD assessment test (CAT) at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  the minimum values is 0 and maximum values is 40, the higher scores mean a worse outcome.
Change from Baseline St George's questionnaire (SGRQ) at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  the minimum values is 0 and maximum values is 100, the higher scores mean a worse outcome.
Change from Baseline Patient Health Questionnaire 9-item (PHQ-9) at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  the minimum values is 0 and maximum values is 27, the higher scores mean a worse outcome.
Change from Baseline Generalized Anxiety Disorder 7-item (GAD-7) at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  the minimum values is 0 and maximum values is 21, the higher scores mean a worse outcome.
Change from Baseline Pittsburgh Sleep Quality Index (PSQI) at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  the minimum values is 0 and maximum values is 21, the higher scores mean a worse outcome.
Change from Baseline Pulmonary Function of FEV1 at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  FEV1
Change from Baseline Pulmonary Function of FVC at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  FVC
Change from Baseline Pulmonary Function of FEV1/FVC at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  FEV1/FVC

OTHER OUTCOMES:
Change from Baseline Body Mass Index (BMI) at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  weight and height will be combined to report BMI in kg/m^2
Change from Baseline Weight in Kilograms at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  weight in kilograms
Change from Baseline Height in Meters at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  height in meters
Change from Waist Circumference in Centimeters at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  waist circumference in centimeters
Change from Hip Circumference in Centimeters at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  hip circumference in centimeters
Change from Waist-Hip Ratio (WHR) at 4, 8, 12 weeks, 6 months and 12 months | baseline and 4, 8, 12 weeks, 6 months and 12 months
  hip and waist circumference in centimeters will be combined to report WHR

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, MD, Study Chair — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang C, Xu J, Yang L, Xu Y, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Huang K, Yao W, Sun T, Shan G, Yang T, Lin Y, Wu S, Zhu J, Wang R, Shi Z, Zhao J, Ye X, Song Y, Wang Q, Zhou Y, Ding L, Yang T, Chen Y, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Chen CS, Wang Z, Zhang H, Bu X, Zhang X, An L, Zhang S, Cao Z, Zhan Q, Yang Y, Cao B, Dai H, Liang L, He J; China Pulmonary Health Study Group. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study): a national cross-sectional study. Lancet. 2018 Apr 28;391(10131):1706-1717. doi: 10.1016/S0140-6736(18)30841-9. Epub 2018 Apr 9. PMID 29650248
- [Result] Alison JA, McKeough ZJ, Johnston K, McNamara RJ, Spencer LM, Jenkins SC, Hill CJ, McDonald VM, Frith P, Cafarella P, Brooke M, Cameron-Tucker HL, Candy S, Cecins N, Chan AS, Dale MT, Dowman LM, Granger C, Halloran S, Jung P, Lee AL, Leung R, Matulick T, Osadnik C, Roberts M, Walsh J, Wootton S, Holland AE; Lung Foundation Australia and the Thoracic Society of Australia and New Zealand. Australian and New Zealand Pulmonary Rehabilitation Guidelines. Respirology. 2017 May;22(4):800-819. doi: 10.1111/resp.13025. Epub 2017 Mar 24. PMID 28339144
- [Result] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Result] Loeckx M, Rabinovich RA, Demeyer H, Louvaris Z, Tanner R, Rubio N, Frei A, De Jong C, Gimeno-Santos E, Rodrigues FM, Buttery SC, Hopkinson NS, Busching G, Strassmann A, Serra I, Vogiatzis I, Garcia-Aymerich J, Polkey MI, Troosters T. Smartphone-Based Physical Activity Telecoaching in Chronic Obstructive Pulmonary Disease: Mixed-Methods Study on Patient Experiences and Lessons for Implementation. JMIR Mhealth Uhealth. 2018 Dec 21;6(12):e200. doi: 10.2196/mhealth.9774. PMID 30578215
- [Result] Storer TW. Exercise in chronic pulmonary disease: resistance exercise prescription. Med Sci Sports Exerc. 2001 Jul;33(7 Suppl):S680-92. doi: 10.1097/00005768-200107001-00006. PMID 11462077